CLINICAL TRIAL: NCT00452673
Title: Phase I Study of Dasatinib (BMS-354825) and Capecitabine for Advanced Breast Cancer
Brief Title: Phase I Study of Dasatinib (BMS-354825) and Capecitabine for Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-004; EUDRACT: 2006-006973-26
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Dasatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50 mg BID dasatinib + 825 mg/m^2 BID capecitabine (Experimental): Twice a day (BID) for 2 weeks of a 3-week cycle
  Interventions: Drug: Dasatinib; Drug: Capecitabine
- 70 mg BID dasatinib + 825 mg/m^2 BID capecitabine (Experimental): BID for 2 weeks of a 3-week cycle
  Interventions: Drug: Dasatinib; Drug: Capecitabine
- 70 mg BID dasatinib + 1000 mg/m^2 BID capecitabine (Experimental): BID for 2 weeks of a 3-week cycle
  Interventions: Drug: Dasatinib; Drug: Capecitabine
- 100 mg QD dasatinib + 1000 mg/m^2 BID capecitabine (Experimental): 2 weeks of a 3-week cycle
  Interventions: Drug: Dasatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 50 mg or 70 mg twice a day (BID), 100 mg once per day (QD). Treatment may continue until disease progression
  Other Names: BMS-354825
Drug: Capecitabine — Tablets, Oral, 660 - 1250 mg/m^2 twice a day (BID). Treatment may continue until disease progression.
  Other Names: Spycel®

SUMMARY:
The purpose of this study is to learn about the safety and efficacy of Dasatinib in combination with Capecitabine for patients with advanced breast cancer, and who have received treatment with a taxane and an anthracycline

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Female with advanced breast cancer previously treated with a taxane and an anthracycline
* No pleural or pericardial effusion
* Not receiving anticoagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (4):
  - City Of Hope National Medical Center, Duarte, California
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - New York Presbyterian Hospital, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington
- Local Institution, Rozzano, Milano, Italy
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Seville

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 Jan 2007 to 30 Oct 2012. Women with advanced breast cancer (ABC) were enrolled.
Pre-assignment Details: 57 enrolled and 52 treated. Reasons for not being treated: 4 no longer met criteria; 1 administrative reason by sponsor. Drug was administered at a reduced dose (gradually escalating at each dose level) during the escalation period and then once a dose for the expansion cohort was identified, additional participants were treated with this dose.
Groups:
- 50 mg Dasatinib + 825 mg/m^2Capecitabine (Dose Escalation): Dose Level 1: 50 milligram (mg) dasatinib oral tablet twice daily (BID) plus 825 mg per meter squared (m^2) capecitabine oral tablet BID. Participants were treated at each dose level (DL) for minimum of 21 days before accrual to the next DL. Rules for dose escalation: If 0 dose level toxicity (DLT) was observed in the first 3 participants in a cohort, the next higher cohort was opened to accrual. If 1 DLT was observed in the first 3 participants in a cohort, then 3 additional participants were studied. If 0 DLT was observed in those 3 (ie, 1 DLT in 6 subjects at the DL), the next higher cohort was opened for accrual. If >=2 DLT was observed in up to 6 subjects, then the maximum tolerated dose (MTD) was exceeded and the next lower DL was defined as the MTD. If 0 DLT was observed in 6 participants in a cohort and the next higher DL exceeded the MTD, then intermediate DLs would be studied. Once the MTD was determined, additional participants were enrolled into that dose group.
- 70 mg Dasatinib + 825 mg/m^2Capecitabine (Dose Escalation): Dose Level 2: 70 mg dasatinib oral tablet BID plus 825 mg/m^2 capecitabine oral tablet BID.
- 70 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Escalation): Dose Level 3: 70 mg dasatinib oral tablet BID plus 1000 mg/m^2 capecitabine oral tablet BID.
- 100 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Escalation): Dose Level 3A: 100 mg dasatinib oral tablet once daily (QD) plus 1000 mg/m^2 capecitabine oral tablet BID. No dose level in this study was identified as the maximum tolerated dose (MDT) but this dose arm (100 mg dasatinib plus 1000 mg/m^2 capecitabine) was selected for expansion in order to provide additional information regarding good tolerance of extended treatment.
- 100 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Expansion): No dose level in this study was identified as the maximum tolerated dose (MDT) but this dose arm (100 mg dasatinib plus 1000 mg/m^2 capecitabine) was selected for the dose expansion period in order to provide additional information regarding good tolerance of extended treatment. An additional 21 participants were treated in this arm in the Dose Expansion Period.
Period: Dose Escalation Period
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine (Dose Escalation) | 70 mg Dasatinib + 825 mg/m^2Capecitabine (Dose Escalation) | 70 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Escalation) | 100 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Escalation) | 100 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Expansion)
Started | 7 | 9 | 6 | 9 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 9 | 6 | 9 | 0
Not completed — Disease Progression | 6 | 6 | 2 | 6 | 0
Not completed — study drug toxicity | 1 | 3 | 3 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Dose Expansion Period
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine (Dose Escalation) | 70 mg Dasatinib + 825 mg/m^2Capecitabine (Dose Escalation) | 70 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Escalation) | 100 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Escalation) | 100 mg Dasatinib + 1000 mg/m^2Capecitabine (Dose Expansion)
Started | 0 | 0 | 0 | 0 | 21 (The last dose level arm in the escalation period was selected for the dose expansion period.)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 21
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 19
Not completed — Other | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 50 mg Dasatinib + 825 mg/m^2Capecitabine: Dose Level 1: 50 milligram (mg) dasatinib oral tablet twice daily (BID) plus 825 mg per meter squared (m^2) capecitabine oral tablet BID. Participants were treated at each dose level (DL) for minimum of 21 days before accrual to the next DL. Rules for dose escalation: If 0 dose level toxicity (DLT) was observed in the first 3 participants in a cohort, the next higher cohort was opened to accrual. If 1 DLT was observed in the first 3 participants in a cohort, then 3 additional participants were studied. If 0 DLT was observed in those 3 (ie, 1 DLT in 6 subjects at the DL), the next higher cohort was opened for accrual. If >=2 DLT was observed in up to 6 subjects, then the maximum tolerated dose (MTD) was exceeded and the next lower DL was defined as the MTD. If 0 DLT was observed in 6 participants in a cohort and the next higher DL exceeded the MTD, then intermediate DLs would be studied. Once the MTD was determined, additional participants were enrolled into that dose group.
- 70 mg Dasatinib + 825 mg/m^2Capecitabine: Dose Level 2: 70 mg dasatinib oral tablet BID plus 825 mg/m^2 capecitabine oral tablet BID.
- 70 mg Dasatinib + 1000 mg/m^2Capecitabine: Dose level 3: 70 mg dasatinib oral tablet BID plus 1000 mg/m^2 capecitabine oral tablet BID.
- 100 mg Dasatinib + 1000 mg/m^2Capecitabine: Dose level 3A: 100 mg dasatinib oral tablet QD plus 1000 mg/m^2 capecitabine oral tablet BID. No dose level in this study was identified as the maximum tolerated dose (MDT) but this dose arm (100 mg dasatinib plus 1000 mg/m^2 capecitabine) was selected for expansion in order to provide additional information regarding good tolerance of extended treatment.
- Total: Total of all reporting groups
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 1000 mg/m^2Capecitabine | 100 mg Dasatinib + 1000 mg/m^2Capecitabine | Total
Number analyzed (Participants) | 7 | 9 | 6 | 30 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.02) | 56.2 (15.52) | 49.5 (10.78) | 54.2 (10.91) | 53.5 (11.56)
Age, Customized [Number; unit: participants]
  < 50 years | 2 | 3 | 3 | 12 | 20
  >= 50 years | 5 | 6 | 3 | 18 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 6 | 30 | 52
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 4 | 17 | 29
  Spain | 2 | 6 | 2 | 11 | 21
  Italy | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities Per Dose Level - Safety Population
Description: Safety was assessed from first dose of study drug through at least 30 days after the last dose, until resolution of drug-related toxicity or when toxicity was deemed irreversible, whichever was longer. An adverse event (AE) was considered a dose limiting toxicity (DLT) if it occurred in the first 21 days and was at least possibly related to study drugs and were: Clinically-evident toxicity of Grade >= 3, or of Grade 2 which required interruption of treatment for >= 7 days (consecutive or non-consecutive); non-hematologic abnormal laboratory value of Grade >= 3, or hematologic toxicity of Grade 4, which persisted 7 days; any grade toxicity which in the judgment of the investigator required a dose reduction or removal from further study therapy.
Time Frame: Day 1 to 30 days post last dose
Population: Safety Population: All participants who received at least one dose of study drug. DLTs: Grade 3 headache, Grade 3 pneumonia, Grade 3 diarrhea in Dosing arms, 1, 2, and 3, respectively. DLTs in dose arm 4: 1 participant with Grade 3 pneumonia and pain and 1 participant with Grade 4 neutropenia and diarrhea plus Grade 3 vomiting and mucositis.
Measure: Number; unit: participants
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 1000 mg/m^2Capecitabine | 100 mg Dasatinib + 1000 mg/m^2Capecitabine
Number analyzed (Participants) | 7 | 9 | 6 | 30
participants | 1 | 1 | 1 | 2

2. Secondary Outcome: Number of Participants With Deaths, Serious Adverse Events, Adverse Events, Adverse Events Leading to Discontinuation and Treatment-related Adverse Events - Safety Population
Description: Adverse events (AEs) were evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Serious AE (SAE)=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: Day 1 up to 30 days post last dose
Population: Safety Population: all participants receiving at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 1000 mg/m^2Capecitabine | 100 mg Dasatinib + 1000 mg/m^2Capecitabine
Number analyzed (Participants) | 7 | 9 | 6 | 30
participants
  Deaths within 30 days of last dose | 0 | 0 | 0 | 0
  Deaths reported beyond 30 days post last dose | 0 | 0 | 0 | 4
  Participants with SAEs | 2 | 2 | 4 | 13
  Participants with Grade 3 - 4 SAEs | 2 | 1 | 4 | 11
  Participants with AEs | 7 | 9 | 6 | 30
  AEs leading to discontinuation of therapy | 2 | 3 | 4 | 4
  Participants with study drug-related AEs | 7 | 9 | 6 | 28

3. Secondary Outcome: Number of Participants With Overall Response to Tumor - Efficacy Evaluable Population
Description: Complete Response (CR): disappearance of all target and non-target lesions, with confirmation at >=4 weeks interval; Partial Response (PR): >= 30% decrease in sum of longest diameter (LDs) of target lesions, taking as reference the baseline sum LD, with confirmation at >= 4 weeks interval. Progressive Disease (PD): Appearance of new lesion(s), or >=20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions. Stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, without unequivocal progression of non-target lesions, after >=6 weeks on study. Radiological tumor assessment by computed tomography (CT) or magnetic resonance imaging (MRI) occurred every 6 weeks. For those patients who were on treatment > 24 weeks, the tumor assessment occurred every 9 weeks.
Time Frame: Day 1 to 30 days post last dose
Population: All participants with at least one measurable lesion at baseline, who received at least one dose of the combination therapy and have at least one on-study tumor assessment or stopped study treatment prior to first assessment, were evaluated. Those who stopped drug prior to tumor assessment for reasons unrelated to disease or drug were excluded.
Measure: Number; unit: participants
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 1000 mg/m^2Capecitabine | 100 mg Dasatinib + 1000 mg/m^2Capecitabine
Number analyzed (Participants) | 4 | 6 | 5 | 25
participants
  Complete Response | 0 | 0 | 0 | 0
  Unconfirmed partial response | 1 | 1 | 1 | 3
  Partial Response | 2 | 1 | 0 | 6
  Stable Disease | 0 | 1 | 2 | 11
  Progressive Disease | 1 | 2 | 2 | 3
  Clinical Progression | 0 | 1 | 0 | 1
  Discontinuation due to study drug toxicity | 0 | 0 | 0 | 1

4. Secondary Outcome: Objective Response Rate (ORR) and Disease Control Rate - Efficacy Evaluable Population
Description: Objective response rate was the percentage of participants, (n/N; number with objective response per Number evaluated) whose best response is either a Complete Response (CR) or a Partial Response (PR). Disease control rate was defined as percentage (n/N) of participants with stable disease greater than (>) 6 months, PR, or CR. Efficacy Evaluable Population: All participants with at least one measurable lesion at baseline, who received at least one dose of combination study drug and have at least one on-study tumor assessment or stopped study treatment prior to first assessment, were evaluated. Those who stop treatment prior to tumor assessment for reasons unrelated to disease or drug were excluded.
Time Frame: Day 1 up to 30 days post last dose
Population: n=number of participants with ORR: 2, 1, 0, 6 in dosing arms 1, 2, 3, and 4, respectively. n= number of participants with Disease control: 3, 2, 2, 14 in dosing arms 1, 2, 3, and 4, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 1000 mg/m^2Capecitabine | 100 mg Dasatinib + 1000 mg/m^2Capecitabine
Number analyzed (Participants) | 4 | 6 | 5 | 25
percentage of participants
  Objective Response Rate | 50.0 [6.76 to 93.24] | 16.67 [0.42 to 64.12] | 0 [NA to NA] — participants=0 so percentage is less than 0 and a Confidence interval is not appropriate. | 24.0 [9.36 to 45.13]
  Disease control rate | 75.0 [19.41 to 99.37] | 33.33 [4.33 to 77.72] | 40.0 [5.27 to 85.34] | 56.00 [34.93 to 75.60]

5. Secondary Outcome: Number of Participants On-Study With Grade 3 - 4 Hematology Laboratory Test Values in Those Participants With a Baseline Laboratory Value of Grade 0 - Safety Population
Description: National Cancer Institute Common terminology criteria (CTC), Version 3 used to assess parameters. Lower limit of normal (LLN). CTC criteria: Absolute neutrophil count (ANC). Leukocytes (White blood cells) Grade (Gr) 1:<LLN to 3.0*10^9/L, Gr 2:<3.0 to 2.0*10^9/L, Gr 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L. ANC Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L. Platelet count Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL. Participants with a baseline hematology lab value of Gr 0 but who had Gr 3 - 4 hematology value while on-study are presented below.
Time Frame: Day 1 up to 30 days post last dose
Population: Safety Population: All participants with at least 1 dose of study drug. N=number of participants with Grade 0 values at baseline in each dosing arm, respectively.
Measure: Number; unit: participants
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 1000 mg/m^2Capecitabine | 100 mg Dasatinib + 1000 mg/m^2Capecitabine
Number analyzed (Participants) | 7 | 9 | 6 | 30
participants
  Leukocytes ( N=7, 9, 5, 29) | 0 | 0 | 0 | 1
  ANC (N=6, 9, 6, 30) | 0 | 0 | 0 | 3
  Platelet Count (N=7, 9, 6, 30) | 0 | 0 | 0 | 1
  Hemoglobin (N=7, 6, 4, 18) | 0 | 0 | 0 | 3

6. Secondary Outcome: Number of Participants On-study With Grade 3 - 4 Chemistry Laboratory Values in Those Participants With a Baseline Laboratory Value of Grade 0 - Safety Population
Description: CTC, Version 3 used to assess parameters. (ULN)=upper limit of normal: (ALT)= alanine transaminase; (AST)=aspartate aminotransferase; (ALP)=alkaline phosphatase. ALT Grade (Gr)1:>ULN to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. AST Gr 1: >ULN to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Total bilirubin Gr 1: >ULN to 1.5*ULN; Gr 2: >1.5 to 3.0*ULN; Gr 3: >3.0 to 10.0*ULN; Gr 4: >10.0*ULN. ALP (U/L) Gr1:>ULN to 2.5*ULN, Gr2:>2.5 to 5.0*ULN, Gr3:>5.0 to 20.0*ULN, Gr4:>20.0*ULN. Albumin (low) Gr 1:<LLN - 3 grams per deciliter (g/dL)to <LLN - 3 g/dL; Gr 2: <3 - 2 g/dL to < 3.0 - 2.0 g/dL; Gr 3: < 2 g/dL to <2 g/L. Participants with a baseline chemistry lab value of Gr 0 but who had Gr 3 - 4 chemistry value while on-study are presented below.
Time Frame: Day 1 to 30 days post last dose
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | 50 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 825 mg/m^2Capecitabine | 70 mg Dasatinib + 1000 mg/m^2Capecitabine | 100 mg Dasatinib + 1000 mg/m^2Capecitabine
Number analyzed (Participants) | 7 | 9 | 6 | 30
participants
  Alkaline Phosphatase (N=4, 6, 5, 21) | 0 | 0 | 0 | 0
  Alanine Aminotransferase (N=6, 9, 6, 25) | 0 | 0 | 0 | 2
  Aspartate Aminotransferase (N=4, 8, 6, 25) | 0 | 0 | 0 | 1
  Total Bilirubin (N=6, 9, 6, 29) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days post last dose.
Groups:
- 50 mg Dasatinib + 825 mg/m^2 Capecitabine: Dose Level 1: 50 milligram (mg) dasatinib oral tablet twice daily (BID) plus 825 mg per meter squared (m^2) capecitabine oral tablet BID. Participants were treated at each dose level (DL) for minimum of 21 days before accrual to the next DL. Rules for dose escalation: If 0 dose level toxicity (DLT) was observed in the first 3 participants in a cohort, the next higher cohort was opened to accrual. If 1 DLT was observed in the first 3 participants in a cohort, then 3 additional participants were studied. If 0 DLT was observed in those 3 (ie, 1 DLT in 6 subjects at the DL), the next higher cohort was opened for accrual. If >=2 DLT was observed in up to 6 subjects, then the maximum tolerated dose (MTD) was exceeded and the next lower DL was defined as the MTD. If 0 DLT was observed in 6 participants in a cohort and the next higher DL exceeded the MTD, then intermediate DLs would be studied. Once the MTD was determined, additional participants were enrolled into that dose group.
- 70 mg Dasatinib + 825 mg/m^2 Capecitabine: Dose Level 2: 70 mg dasatinib oral tablet BID plus 825 mg/m^2 capecitabine oral tablet BID.
- 70 mg Dasatinib + 1000 mg/m^2 Capecitabine: Dose Level 3: 70 mg dasatinib oral tablet BID plus 1000 mg/m^2 capecitabine oral tablet BID.
- 100 mg Dasatinib + 1000 mg/m^2 Capecitabine: Dose Level 3A: 100 mg dasatinib oral tablet once daily (QD) plus 1000 mg/m^2 capecitabine oral tablet BID. No dose level in this study was identified as the maximum tolerated dose (MDT) but this dose arm (100 mg dasatinib plus 1000 mg/m^2 capecitabine) was selected for expansion in order to provide additional information regarding good tolerance of extended treatment.
Arm/Group | 50 mg Dasatinib + 825 mg/m^2 Capecitabine | 70 mg Dasatinib + 825 mg/m^2 Capecitabine | 70 mg Dasatinib + 1000 mg/m^2 Capecitabine | 100 mg Dasatinib + 1000 mg/m^2 Capecitabine
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/9 | 4/6 | 13/30
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 6/6 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Dasatinib + 825 mg/m^2 Capecitabine (N=7) | 70 mg Dasatinib + 825 mg/m^2 Capecitabine (N=9) | 70 mg Dasatinib + 1000 mg/m^2 Capecitabine (N=6) | 100 mg Dasatinib + 1000 mg/m^2 Capecitabine (N=30)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Dasatinib + 825 mg/m^2 Capecitabine (N=7) | 70 mg Dasatinib + 825 mg/m^2 Capecitabine (N=9) | 70 mg Dasatinib + 1000 mg/m^2 Capecitabine (N=6) | 100 mg Dasatinib + 1000 mg/m^2 Capecitabine (N=30)
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 1
Haemoglobin (Investigations) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 6
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 2
Vision blurred (Eye disorders) | 2 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Chills (General disorders) | 2 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 7
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 2 | 12
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 4
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 5
Depression (Psychiatric disorders) | 1 | 2 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 3 | 9
Headache (Nervous system disorders) | 5 | 0 | 3 | 6
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 2
Oedema peripheral (General disorders) | 1 | 0 | 1 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 19
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Aspartate aminotransferase (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 4 | 2 | 12
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 9
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0
Facial neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 2 | 1 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 5
Visual impairment (Eye disorders) | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 7
Chest pain (General disorders) | 1 | 1 | 0 | 2
Diplopia (Eye disorders) | 0 | 0 | 0 | 2
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Hot flush (Vascular disorders) | 1 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 3
Oedema (General disorders) | 0 | 0 | 0 | 2
Pain (General disorders) | 2 | 0 | 1 | 4
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 7
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 1 | 1 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 11
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Neutrophil count (Investigations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 4
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
QRS axis abnormal (Investigations) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 3
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 5
Dizziness (Nervous system disorders) | 1 | 3 | 0 | 5
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 4 | 5 | 3 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 3
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.